CLINICAL TRIAL: NCT00523627
Title: Study of Short-Term Metabolic Adaptation: Prediction of Weight Change and Effects of Macronutrient Manipulations
Brief Title: Effects of Diet Changes on Metabolism
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999907215; 07-DK-N215
Record Dates: First submitted 2007-08-30; First posted 2007-08-31 (Estimated); Last update posted 2026-01-21 (Actual); Status verified 2026-01-16

CONDITIONS: Obesity
Keywords: Energy Expenditure; Adaptive Thermogenesis; Low-protein Overfeeding; Fasting; Weight Gain; Natural History
MeSH Terms: conditions — Obesity; Fasting; Weight Gain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Volunteers with normal glucose regulation: Healthy volunteers with normal glucose regulation

SUMMARY:
This study, conducted at the NIH Clinical Research Unit at the Phoenix Indian Medical Center, will examine how the body s metabolism (energy expenditure) changes when people overeat and when they fast and how different diets (e.g., high-protein or high-fat) affect metabolism. The results may provide information about whether there are mechanisms that make some people more resistant than others to gaining weight when they eat more.

Non-smoking healthy subjects between 18 and 55 years of age who weigh no more than 350 pounds may be eligible for this study. Participants undergo the following procedures:

* Pregnancy test for women of childbearing age.
* Oral glucose tolerance test. For this test, an I.V. line (needle attached to a plastic tube) is inserted into a vein to allow several blood draws without repeated needle sticks. After the first blood sample is drawn, the subject drinks a cola-flavored sugar solution. Five additional blood samples are then drawn over 3 hours.
* Blood test for DNA (genetic) studies related to obesity, diabetes and related medical problems.
* DEXA scan. This test measures body fat. The subject lies on a table while a very small dose of X-rays is passed through the body.
* Respiratory chamber. This test measures how many calories the body burns a day and assesses energy balance between intake and expenditure. Subjects stay in a room with two windows, equipped with a sink, toilet, television and DVD player, desk, chair, telephone and bed for 24 hours. The test is repeated five times during the first 18-day admission and 3 times during the second 13-day admission. For the first two sessions, subjects are fed a diet equal to the amount of energy their body uses. For the next 6 stays they are fed double the amount of calories their body usually uses for 5 of the stays and fast (consume nothing but water and soda without caffeine or calories) during 1 stay. The overfeeding diets may be high or low in protein, normal in protein, or high in fat. Blood tests are done on the day of each respiratory chamber session and a 24-hour urine sample is collected for one day while in the chamber.
* Eating behavior questionnaires.
* Psychological performance tests.

Some participants are asked to volunteer to repeat two of the chamber studies to validate the measurements. The repeat session includes only the fasting and the overfeeding with normal protein content.

All participants are followed at 6 months with blood tests, a DEXA scan, and urine tests (including pregnancy test for women). At annual visits for years 1 through 7, participants have the 6-month tests plus an oral glucose tolerance test.

...

DETAILED DESCRIPTION:
Some people appear to be more resistant than others to gaining weight when they overeat, though they do not increase their physical activity. This may indicate that adaptive mechanisms exist, which lead to wasting as heat part of the excess calories taken in. Such mechanisms exist in rodents including activation of brown fat, a tissue which can also convert calories to heat for warmth. Human studies have provided conflicting results. A pilot study on the relationship of the weight change over time with the changes in the amount of energy an individual uses over 24 hours (energy expenditure, EE) with 48-h overfeeding (OF) and fasting (F) in Pima Indian men has shown that persons with the greatest increase in EE with OF and the smallest decrease in EE with F gained the least weight over time, indicating that the ability to waste more calories when overfed may reduce weight gain. Other studies, however, have not shown this relationship. In addition, it has been proposed that unbalanced diets can help magnify these effects. The aims of this study are to test whether (a) the changes in EE in response to 24-h OF and F predict changes in weight over two years, and (b) high-carbohydrate diets or diets with high or low protein amounts may magnify the metabolic response to 24-h OF compared to normal protein and high-fat diets. 86 volunteers will be evaluated at baseline, 6 months and on a yearly basis for up to 7 years. At baseline, subjects will undergo 8 24-h sessions in a human respiratory chamber to measure EE while on a weight-maintaining diet, and then in random order: fasting, 200% OF on a normal-protein diet, 200% OF on a high fat, low-protein diet, 200% OF on a high-fat, normal-protein diet, 200% OF on a high fat, high protein diet, and 200% OF on a high-carbohydrate, normal-protein diet. Fifteen volunteers will have two additional chambers to try and understand if the source of carbohydrates, i.e. simple sugars versus complex carbohydrates, in a high carbohydrate diet affect metabolism. Thirty volunteers are planned to also undergo 2 positron emission tomography (PET) studies to look at the relationship of brown fat with EE in adult humans. (As of April 2021, we will stop performing the PET scans; 24 volunteers have completed them and we have acquired sufficient data.) Body weight and composition will be measured at each subsequent admission. Hormonal measurements to find determinants of adaptive changes in EE in response to OF and F will also be performed. This study will provide significant insights into possible mechanisms that may help people resist weight gain and obesity.

ELIGIBILITY:
* Inclusion Criteria:
* Age: 18-55 years, to exclude effects of aging on energy expenditure and weight change. For the PET-CT substudy, women will be limited to ages 18-40 years because there is a high likelihood that for women greater than 40 years, their personal physician may recommend an annual routine mammogram, thereby increasing their annual radiation exposure. Men will also be limited to this age range to prevent age discrepancies between men and women for this substudy.
* Premenopausal
* Weight: less than or equal to 450 lb (maximum weight allowed on the DXA scanning tables by the manufacturer).

Exclusion Criteria

* History or clinical manifestation of:
* Current smoking
* Impaired glucose tolerance (IGT), type 1 and type 2 diabetes
* Endocrine disorders, such as Cushing s disease, pituitary disorders, and hypo- and hyperthyroidism
* Pulmonary disorders, including chronic obstructive pulmonary disease, which would limit ability to follow the protocol (investigator judgment)
* Cardiovascular diseases, including coronary heart disease, heart failure, arrhythmias, and peripheral artery disease
* Hypertension, as diagnosed and treated by an outside physician or by sitting blood pressure measurement, using an appropriate cuff, higher than 140/90 mmHg on two or more occasions
* Liver disease, including cirrhosis, active hepatitis B or C, and AST or ALT greater than or equal to 3 times normal
* Renal disease, as defined by serum creatinine concentrations greater than or equal 1.5 mg/dl and/or proteinuria greater than 300 mg/day (200 (Micro)g/min)
* Central nervous system disease, including previous history of cerebrovascular accidents, dementia, and neurodegenerative disorders
* Cancer requiring treatment in the past five years, except for non-melanoma skin cancers or cancers that have clearly been cured or in the opinion of the investigator carry an excellent prognosis (e.g., Stage 1 cervical cancer).
* Infectious disease such as active tuberculosis, HIV (by self-report), chronic coccidiomycoses or other chronic infections that might influence weight.
* Conditions not specifically mentioned above may serve as criteria for exclusion at the discretion of the investigators
* Alcohol and/or drug abuse (more than 3 drinks per day and use of drugs, such as amphetamines, cocaine, heroin, or marijuana).
* Pregnancy or lactation
* For the PET-CT substudy, radiation exposure to the torso for research or medical purposes within the past 12 months
* Positive Urinalysis Drug Screen

Prior to beginning any of the study procedures, all subjects will be fully informed of the aim, nature, and risks of the study prior to giving written informed consent. The study s informed consent will be obtained by a principal or associate investigator, research physician or physician assistant working in the clinical research unit.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Residents of the Phoenix metropolitan area
Sampling Method: Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2008-05-22 (Actual)

PRIMARY OUTCOMES:
Weight, DXA scans, resting metabolic rate, thermic effect of food, energy cost of physical activity, cycle ergometry, core body and distal skin temperature | at baseline visit, 6 month visit, and then annually for up to 7 years
  Changes in body weight and composition in response to changes in energy expenditure
Weight, DXA scans | at baseline visit, 6 month visit, and then annually for up to 7 years
  Changes in body weight and composition in response to overfeeding and fasting diets with high, normal, or low levels of carbohydrates, protein, or fat
Resting metabolic rate, thermic effect of food, energy cost of physical activity, cycle ergometry, core body and distal skin temperature | at baseline visit, 6 month visit, and then annually for up to 7 years
  Changes in energy expenditure in response to overfeeding and fasting diets with high, normal, or low levels of carbohydrates, protein, or fat

SECONDARY OUTCOMES:
Resting metabolic rate, thermic effect of food, energy cost of physical activity, cycle ergometry, FDG-PET and FDG-CT scans, core body and distal skin temperature | at baseline visit, 6 month visit, and then annually for up to 7 years
  Changes in BAT levels in response to cool temperature (16 degrees C), changes in energy expenditure, or changes in diet
Resting metabolic rate, thermic effect of food, energy cost of physical activity, cycle ergometry, core body and distal skin temperature, questionnaires | at baseline visit, 6 month visit, and then annually for up to 7 years
  Predictive value of substrate oxidation in chambers for changes in appetite sensations upon completion of 24 hour respiratory chamber
Resting metabolic rate, thermic effect of food, energy cost of physical activity, cycle ergometry, core body and distal skin temperature | at baseline visit, 6 month visit, and then annually for up to 7 years
  Repeatability of changes in energy expenditure in response to overfeeding and fasting diets with high, normal, or low levels of carbohydrates, protein, or fat
Resting metabolic rate, thermic effect of food, energy cost of physical activity, cycle ergometry, core body and distal skin temperature | at baseline visit, 6 month visit, and then annually for up to 7 years
  Effect of simple sugars and complex carbohydrates during overfeeding on energy expenditure
Resting metabolic rate, thermic effect of food, energy cost of physical activity, cycle ergometry, core body and distal skin temperature | at baseline visit, 6 month visit, and then annually for up to 7 years
  Changes in energy expenditure response to overfeeding in response to thermal insulation of the body core
Hormone values in blood and urine, | at baseline visit, 6 month visit, and then annually for up to 7 years
  Changes in hormones involved in the regulation of energy metabolism in response to overfeeding and fasting diets with high, normal, or low levels of carbohydrates, protein, or fat
Core body and distal skin temperature | at baseline visit, 6 month visit, and then annually for up to 7 years
  Changes in thermic effect of food during overfeeding in response to beta blockade

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Cabeza De Baca, Ph.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- NIDDK, Phoenix, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Trevino-Alvarez AM, Cabeza de Baca T, Stinson EJ, Gluck ME, Chang DC, Piaggi P, Krakoff J. Greater anhedonia scores in healthy individuals are associated with less decline in 24-hour energy expenditure with fasting: Evidence for a link between behavioral traits and spendthrift phenotype. Physiol Behav. 2023 Oct 1;269:114281. doi: 10.1016/j.physbeh.2023.114281. Epub 2023 Jun 24. PMID 37356515
- [Derived] Hollstein T, Basolo A, Unlu Y, Ando T, Walter M, Krakoff J, Piaggi P. Effects of Short-term Fasting on Ghrelin/GH/IGF-1 Axis in Healthy Humans: The Role of Ghrelin in the Thrifty Phenotype. J Clin Endocrinol Metab. 2022 Aug 18;107(9):e3769-e3780. doi: 10.1210/clinem/dgac353. PMID 35678263
- [Derived] Hollstein T, Basolo A, Ando T, Krakoff J, Piaggi P. Reduced adaptive thermogenesis during acute protein-imbalanced overfeeding is a metabolic hallmark of the human thrifty phenotype. Am J Clin Nutr. 2021 Oct 4;114(4):1396-1407. doi: 10.1093/ajcn/nqab209. PMID 34225360
- [Derived] Hollstein T, Basolo A, Ando T, Votruba SB, Walter M, Krakoff J, Piaggi P. Recharacterizing the Metabolic State of Energy Balance in Thrifty and Spendthrift Phenotypes. J Clin Endocrinol Metab. 2020 May 1;105(5):1375-92. doi: 10.1210/clinem/dgaa098. PMID 32118268
- [Derived] Hollstein T, Basolo A, Ando T, Votruba SB, Krakoff J, Piaggi P. Urinary Norepinephrine Is a Metabolic Determinant of 24-Hour Energy Expenditure and Sleeping Metabolic Rate in Adult Humans. J Clin Endocrinol Metab. 2020 Apr 1;105(4):1145-56. doi: 10.1210/clinem/dgaa047. PMID 32002540
- [Derived] Begaye B, Vinales KL, Hollstein T, Ando T, Walter M, Bogardus C, Krakoff J, Piaggi P. Impaired Metabolic Flexibility to High-Fat Overfeeding Predicts Future Weight Gain in Healthy Adults. Diabetes. 2020 Feb;69(2):181-192. doi: 10.2337/db19-0719. Epub 2019 Nov 11. PMID 31712321
- [Derived] Piaggi P. Metabolic Determinants of Weight Gain in Humans. Obesity (Silver Spring). 2019 May;27(5):691-699. doi: 10.1002/oby.22456. PMID 31012296
- [Derived] Vinales KL, Begaye B, Thearle MS, Krakoff J, Piaggi P. Core body temperature, energy expenditure, and epinephrine during fasting, eucaloric feeding, and overfeeding in healthy adult men: evidence for a ceiling effect for human thermogenic response to diet. Metabolism. 2019 May;94:59-68. doi: 10.1016/j.metabol.2019.01.016. Epub 2019 Jan 31. PMID 30710573
- [Derived] Stinson EJ, Graham AL, Thearle MS, Gluck ME, Krakoff J, Piaggi P. Cognitive dietary restraint, disinhibition, and hunger are associated with 24-h energy expenditure. Int J Obes (Lond). 2019 Jul;43(7):1456-1465. doi: 10.1038/s41366-018-0305-9. Epub 2019 Jan 16. PMID 30651576
- [Derived] Begaye B, Piaggi P, Thearle MS, Haskie K, Walter M, Schlogl M, Bonfiglio S, Krakoff J, Vinales KL. Norepinephrine and T4 Are Predictors of Fat Mass Gain in Humans With Cold-Induced Brown Adipose Tissue Activation. J Clin Endocrinol Metab. 2018 Jul 1;103(7):2689-2697. doi: 10.1210/jc.2018-00387. PMID 29788444
- [Derived] Stinson EJ, Krakoff J, Gluck ME. Depressive symptoms and poorer performance on the Stroop Task are associated with weight gain. Physiol Behav. 2018 Mar 15;186:25-30. doi: 10.1016/j.physbeh.2018.01.005. Epub 2018 Jan 9. PMID 29326031
- [Derived] Vinales KL, Schlogl M, Reinhardt M, Thearle MS, Krakoff J, Piaggi P. Cycling Efficiency During Incremental Cycle Ergometry After 24 Hours of Overfeeding or Fasting. Obesity (Silver Spring). 2018 Feb;26(2):368-377. doi: 10.1002/oby.22096. Epub 2017 Dec 25. PMID 29276860
- [Derived] Ibrahim M, Bonfiglio S, Schlogl M, Vinales KL, Piaggi P, Venti C, Walter M, Krakoff J, Thearle MS. Energy Expenditure and Hormone Responses in Humans After Overeating High-Fructose Corn Syrup Versus Whole-Wheat Foods. Obesity (Silver Spring). 2018 Jan;26(1):141-149. doi: 10.1002/oby.22068. Epub 2017 Nov 28. PMID 29193741
- [Derived] Vinales KL, Schlogl M, Piaggi P, Hohenadel M, Graham A, Bonfiglio S, Krakoff J, Thearle MS. The Consistency in Macronutrient Oxidation and the Role for Epinephrine in the Response to Fasting and Overfeeding. J Clin Endocrinol Metab. 2017 Jan 1;102(1):279-289. doi: 10.1210/jc.2016-3006. PMID 27820654
- [Derived] Ibrahim M, Thearle MS, Krakoff J, Gluck ME. Perceived stress and anhedonia predict short-and long-term weight change, respectively, in healthy adults. Eat Behav. 2016 Apr;21:214-9. doi: 10.1016/j.eatbeh.2016.03.009. Epub 2016 Mar 3. PMID 27002703
- [Derived] Schlogl M, Piaggi P, Thiyyagura P, Reiman EM, Chen K, Lutrin C, Krakoff J, Thearle MS. Overfeeding over 24 hours does not activate brown adipose tissue in humans. J Clin Endocrinol Metab. 2013 Dec;98(12):E1956-60. doi: 10.1210/jc.2013-2387. Epub 2013 Sep 30. PMID 24081739
- [Derived] Thearle MS, Pannacciulli N, Bonfiglio S, Pacak K, Krakoff J. Extent and determinants of thermogenic responses to 24 hours of fasting, energy balance, and five different overfeeding diets in humans. J Clin Endocrinol Metab. 2013 Jul;98(7):2791-9. doi: 10.1210/jc.2013-1289. Epub 2013 May 10. PMID 23666976